CLINICAL TRIAL: NCT03666325
Title: Immunotherapy Followed By EGFR Inhibitor In Locally Advanced Or Metastatic Squamous Cell Cancer Of The Skin: Tackling Primary And Secondary Resistance
Brief Title: Immunotherapy +/- EGFR Inhibitor In Advanced/Metastatic cSCC: Tackling Primary And Secondary Resistance
Acronym: I-Tackle
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-Tackle
Record Dates: First submitted 2018-07-16; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Skin Neoplasm
Keywords: metastatic squamous cell cancer of the skin; skin neoplasm; locally advanced squamous cell cancer of the skin; immunotherapy; pembrolizumab; cetuximab
MeSH Terms: conditions — Skin Neoplasms | interventions — pembrolizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab 200 mg, IV infusion on Day 1 of each 3 week cycle. After 3 cycles patient will be evaluated. In case of disease control (SD, PR, CR) the patient will continue to receive pembrolizumab. In case of progression the patient will receive also Cetuximab (250 mg/m2 after loading dose of 400mg/m2 IV infusion every week.
  Interventions: Drug: Pembrolizumab; Drug: Cetuximab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab at 200 mg every 3 weeks for 9 weeks.
  Other Names: Keytruda
Drug: Cetuximab — In case of first progression or no response cetuximab will be added at a weekly dose of 250 mg.
  Other Names: Erbitux

SUMMARY:
Cutaneous Squamous Cell Cancer (Cscc, 25%) and basal cell carcinoma (BCC; 75%) are the major subtypes of non-melanoma skin cancer. Most cSCC arise in the head and neck region because it is frequently exposed to sunlight and its ensuing UV radiation-induced DNA damage, which is the major etiologic factor.

There is an urgent need to identify new therapeutic targets for patients with locally advanced or metastatic squamous Cell Cancer of the skin.

Substantial progress has recently been made in the development of immunotherapy for the treatment of cancer. In particular, the treatment with pembrolizumab alone or in conjunction with an anti epidermal growth factor receptor (EGFR) agent may reverse this condition, so performing radical surgery. Finally, the adjunct of an anti EGFR agent as cetuximab could reverse the primary and secondary resistance to pembrolizumab, with a synergistic effect able to counteract pathway redundancy (i.e. the presence of several concurrent pathways which need to be addressed together) and boosting T cell priming.

Hence, there is rationale to combine cetuximab with pembrolizumab in order to increase its effectiveness.

DETAILED DESCRIPTION:
Cutaneous squamous cell cancers (cSCC) increase in incidence in recent years. Prognosis of these tumors is generally favorable, with most of the patients cured with local therapies, except from a small percentage (less than 10% of the cases) with recurrence not amenable to surgery or radiation or with distant metastasis. There are only limited clinical risk factors able to discriminate an aggressive lesion at its presentation (size > 2cm, perineural invasion (PNI) or beyond subcutaneous tissues). The American Joint Committee on Cancer (AJCC) added aggressive features of cSCC that lead to upstaging the disease and are associated with increased risk of recurrence or metastasis, including invasion of bone, or presence of at least two high-risk factors such as poor differentiation, PNI, invasion greater than 2 mm, occurrence at a high-risk site (i.e., ear or lip), or Clark level greater than or equal to 4.

Untreatable recurrences are most frequently localized in the head and neck area (80% of cases) and they are often disfiguring, while metastasis may involve lymph nodes, lungs, liver or bone. The probability of metastasis in SCC of the skin varies between 2% and 10% depending on the series and on the risk factors considered. Chemotherapy is reserved to cases of recurrence or distant metastasis, with palliative intent. The most commonly used drug combinations are cisplatin-based, in combination with bleomycin, methotrexate, 5-fluorouracil, anthracycline or with cis-retinoic acid and interferon alfa.

However, clinical responses are limited, so underlining the medical need existing with recurrent SCCs of the skin not amenable to local therapy or with metastatic disease.

The role of immunosuppression is well-known in the pathogenesis of skin SCCs; however, only limited evidence exists about the possibility to treat this disease through the restoration of an immune activity against cancer cells. In this regard, there is the need to acquire more information about the expression and the role of the PD-L1:PD1 pathway in skin SCCs, being one of the most attractive in cancer treatment.

In fact, immuno-oncologic agents targeting checkpoint inhibitors such as programmed death receptor-1 (PD-1) or its ligand PD-L1 are very promising new anti-cancer drugs, while efficacy correlates with PD-L1 expression in various tumor types. In order to provide a translational basis for the possible use of PD1/PD-L1 inhibitors in cSCC, Sharper et al examined the expression pattern of PD-L1 in tumor cells and tumor infiltrating leukocytes (TILs) as well as the proportion of CD8+ T- cells and correlated these findings with clinic-pathological characteristics of patients. Utilizing a cut-off ≥ 5%, 10.3% tumors and 42.7% of TILs were PD-L1 positive. The severity of inflammation was positively correlated with PD-L1 expression in both tumor and TILs and PD-L1 expression in tumor cells was associated with the presence of intratumoral CD8+ cells. Additionally, the location of the tumor had an impact on PD- L1 expression: cSCC located in sun-exposed areas (66.2%) showed a higher expression of PD-L1 in TILs compared to cSCC excised in no sun-exposed areas of the body.

Herbst et al. recently showed in multiple cancer types that a response to treatment with a PD- L1 inhibitor was observed especially when PD-L1 was expressed by TILs, therefore the expression of PD-L1 in the majority of TILs in cSCC provides a preclinical rationale for the use of PD-1 inhibitors.

On the other hand, immunohistochemical (IHC) expression of EGFR in skin SCCs is shown to be more than 80%. However, given the paucity of recurrent/metastatic lesions analyzed, only a small amount of data in this setting exists. Primary lesions associated with subsequent metastasis have been shown to more likely overexpress EGFR in comparison with not recurring lesions. Therefore, this pathway represents a potentially valuable target for the treatment of advanced disease. Moreover, HER2 expression is common in skin SCC, being reported with high rates, even if in small studies. Coexpression of EGFR, HER2 and HER3 is present in skin SCCs but not in normal skin and it could be associated with the malignant phenotype.

Anti-EGFR therapy in cSCC has been explored in phase II trials, with cetuximab and panitumumab in unresectable or metastatic setting, with gefitinib in potentially curable disease and in other case reports.

EGFR-TKI gefitinib was shown to reduce the expression of PD-L1 in both EGFR-TKIs sensitive and acquired resistant non-small cell lung cancer in vitro and in vivo, so providing a novel anti-tumor mechanism for the combination of EGFR-TKIs and immunotherapy.

Being the responses to cetuximab alone are limited and not durable, there is the need to enhance response rate and secondarily duration of responses. There are suggestions for a possible role of anti-EGFR agent in tackling resistance to checkpoint inhibitors. In fact, suppression of EGFR signalling decreases PD-L1 overexpression on tumoral cells (possible mechanism of resistance to immunotherapy), so reducing the immune escape process. Moreover, activation of EGFR pathway is involved in suppressing the immune response through activation of Tregs or reducing the level of T cell chemoattractants.

Recently, an anti-PD-1 monoclonal antibody employed in patients with unresectable locally advanced or metastatic cSCC showed activity and a tolerable profile of toxicity.

After confirmation of inclusion/exclusion criteria, the patient will be treated with pembrolizumab 200 mg every 3 weeks.

First evaluation: After 9 weeks since treatment start the patient will be evaluated clinically and radiologically, if indicated.

In case of disease control (SD/PR/CR), the patient will continue to receive pembrolizumab alone and after 6 weeks will be evaluated clinically and radiologically, if indicated.

In case of disease progression at the first evaluation, in order to avoid disease pseudo-progression, the patient will repeat an evaluation (confirmatory) after at least 4 weeks; if PD confirmed, then the patient will receive cetuximab (400 mg/sm loading dose, then 250 mg/sm day 1,8 and 15 of a 3-week schedule) in addition to pembrolizumab.

Second and following evaluations: After the first evaluation, every restaging will be performed every 6 weeks.

In case of disease response (PR/CR), the patient will continue to receive pembrolizumab alone.

In case of stable disease or progression, the patient will repeat an evaluation after at least 4 weeks (confirmatory); in case of confirmed stability or PD, the patient will receive cetuximab (400 mg/sm loading dose, then 250 mg/sm day 1,8 of a 3-week schedule) in addition to pembrolizumab, in order to reverse the primary lack of response to the immunotherapeutic drug.

In case of progression after an initial disease response, the patient will receive cetuximab (400 mg/sm loading dose, then 250 mg/sm day 1,8, 15 of a 3-week schedule) in addition to pembrolizumab, in order to reverse the acquired resistance to the immunotherapeutic drug.

After 6 weeks of combination treatment (pembrolizumab + cetuximab) a first clinical/radiological assessment will be performed. In case of lack of response (PR or CR), another assessment will be performed within 4 weeks. In case of confirmed lack of response during the combination treatment the patient will be permanently discontinued from study, as the balance of possible treatment toxicities against its lack of efficacy is no more favorable.

Evaluation will be conducted according to the ir-RECIST Partial response will be considered at any time according to ir-RECIST with a reduction ≥50% in tumor burden compared with the first assessment at study entry for each treatment schedule. The first 6 patients treated with the combination of pembrolizumab and cetuximab will be treated within a safety run-in cohort.

The safety run-in cohort will include 6 subjects treated with 250 mg/sm (after loading dose 400 mg/sm) IV infusion of weekly cetuximab plus standard-dose pembrolizumab. These first 6 patients will be followed for 4 weeks for dose limiting toxicities (DLT) before enrolling additional patients.

If a DLT will be observed in no more than 1 of 6 patients, the trial will continue with enrolling subjects to the remainder of the phase II portion of the study. Otherwise, 6 additional patients will be enrolled at dose level -1 (200 mg/sm).

If no more than one DLT will be observed, then phase II will enroll patients at dose level -1 (200 mg) for the total expected number of accrual.

If a DLT will be observed in more than 1 of 6 patients, 6 additional patients will be enrolled at dose level -2 (150 mg).

If no more than one DLT will be observed with this dose level, then phase II will enroll patients at dose level -2 (150 mg) for the total expected number of accrual. Otherwise the combination of the 2 drugs will be considered unfeasible in such a disease population.

To consolidate these safety data, after 6 patients will have completed treatment at the specific dose without more than one DLT, other 6 patients will be analyzed for safety purpose, without the need to stop enrollment. In case 3 or more DLTs will globally happen in the 12 treated patients, then the trial will continue to enroll 6 additional patients at the inferior dose level with the above reported rules.

Primary Objective(s) & Hypothesis(es):

(1) Objective: Increase in cumulative response rate (PR + CR) obtained by single agent or by combination strategy (pembrolizumab alone or with pembrolizumab + EGFR inhibiting agent) in respect to monotherapy with anti-EGFR agent.

Hypothesis: this approach will be considered effective if the cumulative response rate is at least 45%, with an increase of 17% with respect to previous study with cetuximab in the same setting of disease, in which a response rate of 28% was shown.

Secondary Objective(s) & Hypothesis(es)

* Compliance to the treatment and safety
* Disease control (SD + PR + CR) as best response obtained by single agent or by combination
* Progression-Free Survival (PFS) and Overall Survival (OS)
* Percentage of patients initially not considered for surgery due to difficulty to obtain a curative treatment that undergo surgery after the treatment (pembrolizumab alone or pembrolizumab + anti EGFR agent)
* Reversal of acquired resistance to pembrolizumab obtained through the addition of cetuximab (percentage of responding patients after cetuximab adjunct) 4.3 Exploratory Objective Translational research (TR): In skin cancers performing paired biopsies is relatively easy.

Patients will be asked to consent to analysis of tissue and to receive additional biopsies at time of anti EGFR agent introduction; if possible, another biopsy at time of combined therapy resistance will be acquired.

TR includes: - evaluation of PD-L1 expression in skin SCC and of PD1 on CD8 T cells at baseline , - evaluation of PD-L1 and PD1 modulation during treatment, -evaluation of PDL-1 and PD-1 in TILs at the baseline and during treatment.

* evaluation of the presence of HPV genotype on tumor sample through viral DNA and RNA detection by PCR.
* evaluation of pharmacodynamic changes of potential markers in course of therapy, and their association with response to treatment.

Moreover, the study will involve a multi-omic approach with analysis of gene-expression, miRNA, methylation and CGH profiling, completed by next generation "amplicon sequencing", by means of Ion Torrent, detecting with high sensitivity mutations and polymorphisms of biomarkers associated with prognosis and with response to the whole treatment.

Initially, a bio-banking of FFPE (formalin-fixed paraffin-embedded ) tissues and of blood will be performed, as this part of the analysis has not been funded yet. A separate consent will be requested for additional biopsies and for bio-banking.

The pre-pembrolizumab and pre-cetuximab biopsies will be compared in order to evaluate the changes in microenvironment and tumoral pharmacodynamic markers.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent/assent for the trial.
* 18 years of age.
* Histological diagnosis of squamous cell carcinoma of the skin not amenable to surgical treatment and to radiation with curative purposes or with clinical contraindication to surgery and radiation.
* Have metastatic disease
* Have measurable disease based on RECIST 1.1.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Demonstrate adequate hematological, renal and hepatic organ function as defined in the study protocol.
* Women of childbearing potential should have a negative pregnancy within 72 hours prior to receiving the first dose of study medication.
* Women of childbearing potential must be willing to use an adequate method of contraception as outlined in the study protocol4
* Men of childbearing potential must be willing to use an adequate method of contraception as outlined in the study protocol

Exclusion Criteria:

* Current or past participation participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Previous treatment with anti-EGFR agent
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (prednisone equivalent dose > 10 mg per day) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to the trials drugs or their excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (≤ Grade 1 or at baseline) from adverse events.
* Has a known additional malignancy that is progressing or requires active treatment.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has active autoimmune disease that has required systemic treatment in the past 2 years.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with participation, or is not in the best interest of the subject.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has previously received an organ transplant
* Has previously received bone marrow transplantation
* Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative response rate | 15 patients will be enrolled. The first evaluation will take place when the last completes three 21-day cycles of Pembrolizumab+/-cetuximab. If we don't observe at least 5 responses (PR/CR), we will stop the recruitment and reject the hypothesis.
  Increase in cumulative response rate (PR + CR) obtained by single agent or by combination strategy (pembrolizumab alone or with pembrolizumab + EGFR inhibiting agent) in respect to monotherapy with anti-EGFR agent.

SECONDARY OUTCOMES:
Compliance and safety | Treatment emergent adverse events will be measured throughout the study treatment (at each 21-days cycle.).
  Treatment safety will be evaluated by the frequency, type and severity of adverse events, graded according to NCI-CTCAE v.4.03
Best response | After first evaluation (after 9 weeks), every restaging will be performed every 6 weeks
  Disease control (SD + PR + CR) as best response obtained by single agent or by combination
PFS | through study completion, an average of 4 years. PFS calculated in each patient as the time from the date of treatment start to the date of first progression or death, whichever comes first
  Progression free survival
OS | through study completion, an average of 4 years. OS, calculated for each patient as the time from the date of treatment start to the date of death.
  Overall survival
Proportion of patients undergoing surgery | Through study completion an average of 4 years
  Percentage of patients initially not considered for surgery due to difficulty to obtain a curative treatment that undergo surgery after the treatment (pembrolizumab alone or pembrolizumab + anti EGFR agent)
percentage of responding patients | Through study completion, an average of 4 years
  Reversal of acquired resistance to pembrolizumab obtained through the addition of cetuximab (percentage of responding patients)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bossi, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (7):
- Italy (7):
  - ASST Spedali Civili di Brescia, Brescia, BS
  - Azienda Ospedaliero Universitaria Careggi, Florence, FI
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI
  - Istituto Europeo di Oncologia, Milan, MI
  - Ospedale di Circolo e Fondazione Macchi, Varese, VA
  - Istituto IRCCS AOU S. Martino, Genova
  - Istituto Nazionale Tumori - Fondazione IRCCS "G. Pascale", Napoli

IPD SHARING:
Plan to Share IPD: No